CLINICAL TRIAL: NCT07407101
Title: Optimization of Autologous Serum Eye Drops: Study of Filtration on Active Molecule Concentration in Patients With Dry Eye Disease (IFilCoSA)
Brief Title: Impact of Filtration on Autologous Serum Eye Drops
Acronym: IFILCOSA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 87RI25_003 (IFILCOSA)
Record Dates: First submitted 2026-01-19; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Dry Eye Syndrome (DES)
Keywords: Dry Eye Syndrome; Autologous serum; eye drops; filtration; pilot project; active molecules of autologous serum; TGF β; IGF 1; EGF; fibronectin; vitamin A
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Insulin-Like Growth Factor I; Epidermal Growth Factor; Fibronectins; Vitamin A

STUDY DESIGN:
Intervention Model Description: Pilot study, descriptive study
Masking Description: The biological analyses are carried out blindly
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Serum (Experimental): analyse sera
  Interventions: Biological: Serum dosage of TGF-β, IGF-1, EGF, Fibronectin and Vitamin A

INTERVENTIONS:
Biological: Serum dosage of TGF-β, IGF-1, EGF, Fibronectin and Vitamin A — Dosage of active molecules of autologous serum: TGF β, IGF 1, EGF, fibronectin and vitamin A

SUMMARY:
Dry eye disease accounts for nearly 25% of ophthalmology consultations, making it a commonly encountered condition. When conventional treatments fail autologous serum in the form of eye drops, have been proposed as a therapeutic option. With the aim of standardizing the preparation of autologous serum eye drops in France, the main objective is to describe the absolute and relative differences (before and after filtration) in the concentrations of active molecules in the autologous serum of patients suffering from severe dry eye disease.

DETAILED DESCRIPTION:
Sterility, which is a mandatory specification for eye drops, represents a critcial step in their manufacturing process. A review of the literature shows that 62% of articles (n=42) addressing the manufacturing process of autologous serum eye drops do not include a filtration step. Among those reporting filtration, slightly over 9% do not specify the porosity used, 4.8% use filters with a porosity of 0.45µm (clarifying filtration), and slightly over 23% use filters with a porosity ≤ 0.22µm ( sterilizing filtration). Several molecules present in autologous serum have been described in the literature, but five are widely recognized as the main contributors to its therapeutic efficacy: EGF, TGF-ß, IGF-1, Fibronectin, and Vitamin A. The impact of sterilizing filtration on the concentrations of thesemolecules in the final serum used for eye drop preparation therefore warrants investigation. Ten patients will be recruited from the ophthalmology department. A pre-screening phase will be conducted to identify eligible patients and propose the study participation. A dedicated follow-up consultation will be organized for inclusion. Serological tests will be performed on the blood samples of eligible patients. Only patients with negative serology for HIV, HBV, HCV and Treponema pallidum will be included. Their serum will be processed, at the Pharmaceutical Preparations Unit, to produce multiple aliquots following coagulation and centrifugation, with subsequentfiltration using 2 different filter materials, with 2 different porosities, or no filtration. These aliquots will then be sent to the Biochemistry department and Pharmacology department for the quantitative analysis of molecules of interest.

ELIGIBILITY:
Inclusion Criteria:

* adult patients
* patients covered by health insurance
* patients managed by the Ophtalmology Department of the University Hospital of Limoges
* patients diagnosed with dry eyes syndrome, who have not responded to conventionnal treatments
* free, informed, written and signed consent

Exclusion Criteria:

* person incapable of consent
* legal guardianship or wardship
* patient who does not wish to know the results of serological tests

Secondary exclusion criteria:

- a positive serology for at least of of the following agents (HIV, HCV, HBV or syphilis)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2026-04-30 (Estimated); Primary Completion 2027-04-29 (Estimated); Study Completion 2027-04-29 (Estimated)

PRIMARY OUTCOMES:
Differences in concentrations of active molecules | At the inclusion
  Absolute and relative differences in concentrations, before/after filtration (clarifying or sterilizing, and using polyethersulfone or cellulose acetate), of the following active molecules: EGF, TGF-ß, IGF-1, Fibronectin, and Vitamin A.

SECONDARY OUTCOMES:
Concentration of active molecules | At the inclusion
  The impact of filtration is considered significant if the relative decrease in concentrations following filtration is ≥ 7,5% given the galenic form.
Physiological parameters of patients to graduate chronical dry eye disease | At the inclusion
  Symptoms; therapeutic management of dry eye syndrom; diagnostic tests performed and contributory elements to the diagnosis: slit lamp examination and standard Oxford scale for fluorecein staining; graduate in severe intermediate and early stages
OSDI quality of life questionnary | At the inclusion
Description of the concentrations of active molecules in the serum before filtration. | At the inclusion
  Average value of the concentrations measured in duplicate for each active compound in a given patient.
Description of the proposed patient pathway and manufacturing process. | From the inclusion to the end of results 7 days later
  Record the time taken for each step of the process, from sample collection to the availability of the assay results, as well as any incidents that occurred or comments from the personnel involved at each stage.

CONTACTS AND LOCATIONS:
Overall Officials: Maxime Rocher, Dr, Principal Investigator — University Hospital, Limoges
Locations (1):
- CHU Limoges, Limoges, France

IPD SHARING:
Plan to Share IPD: Undecided